CLINICAL TRIAL: NCT01557413
Title: Randomised Study Between Intramedullary Locking Nails and Locking Plates for Treatment of Proximal Humerus Fractures in Patients After 40-year-old
Brief Title: Randomised Study Between Intramedullary Locking Nails and Locking Plates for Treatment of Proximal Humerus Fractures
Acronym: HUMERUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOO269-32
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Proximal Humerus Fractures
Keywords: Humerus; fracture; nail; plate; tuberosity
MeSH Terms: conditions — Fractures, Bone | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramedullary nail (Experimental): Intramedullary nail
  Interventions: Procedure: Intramedullary nail
- Locked plate (Experimental): Locked plate
  Interventions: Procedure: Locked plate

INTERVENTIONS:
Procedure: Intramedullary nail — the fracture was reduced and fix by an intramedullary humeral nail (Multilock, SYNTHES, Switzerland) using an open surgery. An anterolateral approach will be performed, the patient sit in beach chair position under general anesthesia. If required additional sutures will be authorized to fix the tuberosities.
  Other Names: SURFIX, Integra
  Arms: Intramedullary nail
Procedure: Locked plate — the fracture was reduced and fix by a locking plate using an open surgery (SURFIX, Integra, France). A deltopectoral approach will be performed, the patient sit in beach position under general anesthesia. If required, additional sutures will be authorized to fix the tuberosities.
  Other Names: Multilock, SYNTHES
  Arms: Locked plate

SUMMARY:
Primary purpose of this study was to compare functional outcomes after displaced and proximal humerus fracture between nails and locked plates.

The hypothesis is that intramedullary nails provides satisfactory fixation and functional outcome compared to locked plate.

DETAILED DESCRIPTION:
: Proximal humerus fractures have a higher occurrence in elderly patients and therefore represent a public health problem.

Prognosis depends on greater and lesser tuberosity status, where rotator tendons of the shoulder have their insertion site.

Surgical treatment is recommended in case of tuberosities displacement. Goals are their anatomic reduction and stable primary fixation that will allow good bone healing and early mobilization. It has been demonstrated that an extended immobilization can result in stiffness by capsular retraction. On the contrary a too early mobilization can lead to secondary displacement of tuberosities and malunion.

These sequelae can be responsible for real disability when occuring in active patients, in particular when dominant limb is affected.

Internal fixation by locking intramedullary nails is currently the first choice technique because less invasive. However it doesn't always provide a good bone fixation, leading to tuberosities displacement or longer immobilization that decrease shoulder function prognosis. Locking plates represent a good alternative to avoid these complications by offering a better fixation of tuberosities in osteoporotic bone.

Though there is no existing randomised study comparing these techniques regarding functional outcomes, complications rates, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patients between 40 and 85-years-old, who didn't expressed opposition to inclusion, with type III or IV displaced CEPHALOTUBEROSITY fracture( classification of Neer and DUPARC).

Exclusion Criteria:

* CEPHALOTUBEROSITY fractures type IV - CT4 will not be included because it can correspond to posterior or anterior fracture-dislocation of humeral head and therefore be associated to very high risk level of avascular necrosis . In this case a surgical treatment by arthroplasty is recommended.

Dislocated fracture Patient who express opposition to inclusion polytrauma

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Constant and MURLEY Score | 12 months
  comparison of shoulder function outcome between 2 groups using Constant- Murley score after 12 months( mobility, function, pain and strength)

SECONDARY OUTCOMES:
Quick Dash, complication (mal union, necrosis, infection) | 6 and 18 months
  comparison of Constant-Murley score after 6 and 18 months, comparison of complications rates and patients satisfaction( DASH and STT scores).
  Those criteriae will be analysed on global groups and for each Neer and Duparc classification type fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boyer, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard 46, rue Henri-Huchard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196